CLINICAL TRIAL: NCT06461507
Title: Effects of Jandas's Approach With and Without Post Isometric Relaxation Technique on Pain, Muscle Flexibility, Functional Disability in Patients With Posterior Lower Crossed Syndrome
Brief Title: Comparative Effects of Jandas's Approach With and Without Post Isometric Relaxation Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0194 Nimra
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: PELVIS Syndrome
Keywords: disability; pain; flexibility
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Muscle Energy Technique (METs) (Experimental): ▪ Apply METs to the iliopsoas muscle by instructing the patient to do hip flexion and resist movement by pushing their leg down towards the table, activating their iliopsoas muscle. (This contraction is known as an isometric contraction). Maintain the isometric contraction for approximately 5-10 seconds, encouraging the patient to exert maximal effort. After the contraction, relax the patient's leg as they exhale, and take the muscle to its new, slightly increased, passive range of motion.
  Interventions: Other: Janda's Approach
- Group B: Janda's Approach (Active Comparator): For tightened structures stretching, use the Iliopsoas stretch and the Erector spinae stretch (5 repetitions of stretching with 30-s hold for each muscle) For Strengthening Weakened Structures: Glute bridge, Abdominal crunch (10 repetitions of each)
  Interventions: Other: Janda's Approach

INTERVENTIONS:
Other: Janda's Approach — For Tightened Structures Stretching applied toIliopsoas and Erector spinal muscles (5 repetitions of stretching with 30-s hold for each muscle). For Strengthening of Weakened Structures; Glute bridge and Abdominal crunch(10 repetitions of each).

SUMMARY:
Posterior lower crossed syndrome is a perplexing puzzle of muscular imbalance, manifests as an intricate interplay between weakened glutes and tight flexors. The aim of the study will be to determine the effects of Jandas's approach with and without post-isometric relaxation technique on pain, muscle flexibility, and functional disability in patients with the posterior lower crossed syndrome.

DETAILED DESCRIPTION:
A Randomized Controlled Trial will be conducted at physical therapy department of Rabia Welfare Hospital Lahore, FMH Physiotherapy Clinic Lahore and Shafaeen Physiotherapy Clinic Lahore through convenient sampling technique on 30 patients which will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will be treated with janda's approach and Group B will be treated with combination of post isometric relaxation technique for Illiopsoas and janda's approach at the frequency of 3 sets with 10 repetitions and twice a week. Outcome measures will be conducted through pain,muscle flexibility, pelvic tilt and disability questionnaire after 4 weeks. Data will be analysed using SPSS software version 25.After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or nonparametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age:20-60 years
* Gender: Both males and females
* NPRS (Numerical Pain Rating Scale): < 7
* Positive Finger to Floor Test : > 48cm in males, >50cm for females
* Positive Modified Thomas Test: greater than zero
* Patients with anterior pelvic tilt

Exclusion Criteria:

* Preexisting spinal pathology
* Congenital abnormality
* Neurological deficits,
* Recent spinal or lower-limb trauma or surgery
* Spasm of the trunk or lower-limb muscles
* Lower-limb radiculopathy
* Pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Numerical pain rating scale (NPRS) | upto 4 weeks
  o Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Finger to floor test -Muscle flexibility test | upto 4 weeks
  * The patient is asked to bend forward and attempt to reach for the floor with their fingertips.
  * The physical therapist then measures the distance between the patient's right long finger and the floor using a standard measuring tape
  * Ask the client whether pain, stiffness or both limit the movement(Fingertips to floor (FTF) test).
  * If the FTF test is limited by pain, the location and pain score out of 10 should be documented.
  * If the FTF test is 0 cm or the patient is able to place their palms to the floor with no pain, a different outcome measure should be considered.
Modified Thomas Test- Muscle flexibility test | upto 4 weeks
  * Have the patient lie supine on a firm surface, with their legs straight.
  * Place your hand under the patient's lower back to maintain a neutral spine.
  * Slowly flex the patient's hip, bringing their knee towards their chest, until their thigh is perpendicular to the table.
  * Assist the patient in flexing their hip further, keeping their knee bent at a 90-degree angle.
  * Measure the angle between the patient's thigh and the table using a goniometer or inclinometer.
  * Compare the measurement to the normal range (usually around 15-20 degrees) to determine if there is a restriction in iliopsoas flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Nimra Azhar, MSPT*, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Shafeen medical complex Punjab Pakistan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Key J. 'The core': understanding it, and retraining its dysfunction. J Bodyw Mov Ther. 2013 Oct;17(4):541-59. doi: 10.1016/j.jbmt.2013.03.012. Epub 2013 Jun 28. PMID 24139017
- [Background] Roberts JM, Wilson K. Effect of stretching duration on active and passive range of motion in the lower extremity. Br J Sports Med. 1999 Aug;33(4):259-63. doi: 10.1136/bjsm.33.4.259. PMID 10450481
- [Background] Kale, S. S. and S. Gijare (2019).
- [Background] Ishida H, Hirose R, Watanabe S. Comparison of changes in the contraction of the lateral abdominal muscles between the abdominal drawing-in maneuver and breathe held at the maximum expiratory level. Man Ther. 2012 Oct;17(5):427-31. doi: 10.1016/j.math.2012.04.006. Epub 2012 May 16. PMID 22595657
- [Background] Esakowitz, A. (2014). The effect of muscle energy technique versus chiropractic adjustive therapy in the treatment of chronic low back pain with lower cross syndrome, University of Johannesburg (South Africa).
- [Background] Janda, V. (1987).